CLINICAL TRIAL: NCT05139472
Title: Impact of Empagliflozin on Functional Capacity in Heart Failure with Preserved Ejection Fraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, James MacNamara, Assistant Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 2018-0311
Record Dates: First submitted 2021-11-10; First posted 2021-12-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure with Preserved Ejection Fraction; Heart Failure, Diastolic; Diabetes Mellitus
Keywords: Exercise; Invasive Exercise Testing; SGLT-2 Inhibitors
MeSH Terms: conditions — Heart Failure, Diastolic; Diabetes Mellitus; Motor Activity | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Single arm, open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): This arm of the study will take 10 mg empagliflozin daily for 12 weeks
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Daily Empagliflozin

SUMMARY:
Sodium-Glucose Cotransporter-2 (SGLT-2) inhibitors generally and empagliflozin specifically have shown cardiovascular benefits in patients with heart failure (HF), but the underlying mechanisms remain unclear. Empagliflozin use resulted in lower pulmonary artery diastolic pressures in patients with HF, suggesting a beneficial diuretic effect. Other potential mechanisms include increased blood volume, decreased blood pressure, and changes in sympathetic and neuro-hormonal activation.

This study is a single-arm, open label, prospective interventional study of 8 subjects with heart failure with preserved ejection fraction (HFpEF). Before and after 12 weeks of daily empagliflozin, participants with undergo comprehensive invasive exercise testing with a right heart catheter. Our goal is to evaluate the effects of empagliflozin on fitness, assessed by peak VO2, and peak left ventricular filling pressure, assessed by pulmonary capillary pressure at peak exercise.

DETAILED DESCRIPTION:
This is a single-arm, open label, pilot study of 8 subjects with HFpEF. The subjects will undergo screening tests (exercise stress echo and blood work) to evaluate for potential exclusion criteria and provide familiarization to the exercise protocol. Those included will undergo an echocardiogram and invasive cardiopulmonary exercise test. This involves placement of a right heart catheter in the pulmonary artery and undergoing seated, upright exercise. During the exercise test, the subject's oxygen uptake (VO2), intra-cardiac pressures (right atrial pressure, pulmonary capillary wedge pressure) and cardiac output (Qc) will be measured. The subject will take a dose of empagliflozin in the lab and wait for at least 60 minutes. They will repeat a shortened version of the exercise test in the afternoon. After baseline testing, each subject will take 10mg empagliflozin daily for 12 weeks. They will have repeat blood work (specific electrolytes and renal function) 30 days after starting medication to screen for renal injury. After 12 weeks, they will return for another invasive cardiopulmonary exercise test and echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* adults ages 50-85
* clinical heart failure
* ejection fraction > 50%

Exclusion Criteria:

* previous hypersensitivity or adverse reaction to SGLT-2 inhibitors
* currently treated with SGLT-2 inhibitor
* current or prior ejection fraction <50%
* chronic kidney disease with glomerular filtration rate < 45 ml/kg/min
* unstable coronary artery disease
* significant arrhythmia
* BMI >55 kg/m2
* inability to exercise.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Peak Oxygen Uptake | 12 weeks
  Peak VO2 measured on maximal exercise test
Peak Pulmonary Capillary Wedge Pressure (PCWP) | 12 weeks
  Peak PCWP, measured at end-expiration, at the end of maximal exercise test

SECONDARY OUTCOMES:
Primary Endpoints after single dose of empagliflozin | 1 hour
  Peak VO2 and peak PCWP will be measured after a single dose of empagliflozin
Cardiac Output at Rest and During Exercise | 12 weeks
Stroke Volume at Rest and During Exercise | 12 weeks
Right Atrial Pressure at Rest and During Exercise | 12 weeks
Pulmonary Capillary Wedge Pressure at Rest and During Submaximal Exercise | 12 weeks
Left ventricular volumes at rest and during submaximal exercise | 12 weeks
  Measured by echocardiography
Hemoglobin mass, plasma volume, total blood volume | 12 weeks
  Measured by Carbon Monoxide Rebreathe
Diastolic parameters at rest and during submaximal exercise | 12 weeks
  Measured by echocardiography
6 minute walk time | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Institute for Exercise and Environmental Medicine, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
De-identified data may be made available upon reasonable request